CLINICAL TRIAL: NCT02160756
Title: A Single-Dose, Open-Label, Randomized, Parallel-Group Study to Assess the Relative Bioavailability of 3 Tablet Formulations of JNJ-56021927 With Respect to the Capsule Formulation of JNJ-56021927 Under Fasted Conditions in Healthy Male Subjects
Brief Title: Bioavailability Study of 3 Tablet Formulations vs. Capsule Formulation of JNJ-56021927 in Fasting Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aragon Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR104824; 56021927PCR1011 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2014-06-09; First posted 2014-06-11 (Estimated); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Healthy
Keywords: Healthy; JNJ-56021927; JNJ-56142060; ARN-509
MeSH Terms: interventions — apalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Treatment A (Active Comparator): Single oral dose of JNJ-56021927 240 milligram (mg) softgel capsule on Day 1.
  Interventions: Drug: JNJ-56021927 Softgel Capsule
- Treatment B (Experimental): Single oral dose of JNJ-56021927 240 mg Tablet Formulation 1 on Day 1.
  Interventions: Drug: JNJ-56021927 Tablet Formulation 1
- Treatment C (Experimental): Single oral dose of JNJ-56021927 240 mg Tablet Formulation 2 on Day 1.
  Interventions: Drug: JNJ-56021927 Tablet Formulation 2
- Treatment D (Experimental): Single oral dose of JNJ-56021927 240 mg Tablet Formulation 3 on Day 1.
  Interventions: Drug: JNJ-56021927 Tablet Formulation 3

INTERVENTIONS:
Drug: JNJ-56021927 Softgel Capsule — Single oral dose of JNJ-56021927 240 mg softgel capsule on Day 1.
  Other Names: ARN-509
  Arms: Treatment A
Drug: JNJ-56021927 Tablet Formulation 1 — Single oral dose of JNJ-56021927 240 mg Tablet Formulation 1 on Day 1.
  Arms: Treatment B
Drug: JNJ-56021927 Tablet Formulation 2 — Single oral dose of JNJ-56021927 240 mg Tablet Formulation 2 on Day 1.
  Arms: Treatment C
Drug: JNJ-56021927 Tablet Formulation 3 — Single oral dose of JNJ-56021927 240 mg Tablet Formulation 3 on Day 1.
  Arms: Treatment D

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics (PK - the study of the way a drug enters and leaves the blood and tissues over time) and relative bioavailability (the extent to which a drug or other substance becomes available to the body) of JNJ-56021927, when administered as 3 tablet formulations (test) compared with JNJ-54781532 softgel capsule formulation (reference) in healthy male participants under fasted conditions at a single dose of 240 milligram (mg).

DETAILED DESCRIPTION:
This is a randomized (study medication assigned to participants by chance), open-label (all people know the identity of the intervention), single-center, 4-treatment, parallel design (a medical research study comparing the response in two or more groups of participants receiving different interventions) study of a single dose of 240 mg JNJ-56021927. The duration of study will be approximately of 78 days per participant. The study consists of 3 parts: Screening phase (that is, 21 days before study commences on Day 1); Open-label Treatment phase (consists of 4 parallel single-dose treatments); and End-of-Study (completion of the Hour 1344 PK sampling on Day 57, or upon early withdrawal). All the eligible participants will be randomly assigned to 1 of the 4 possible treatments: Treatment A (240 mg dose as softgel capsule); Treatment B (240 mg dose as Tablet Formulation 1); Treatment C (240 mg dose as Tablet Formulation 2); or Treatment D (240 mg dose as Tablet Formulation 3). Participants will fast overnight from food and fluids (excluding non-carbonated water) for at least 10 hours before study drug administration on Day 1. Blood samples will be collected pre-dose and over 1,344 hours (Day 57) after dosing for the determination of JNJ-56021927 concentration and its active metabolite. Relative bioavailability of 3 tablet formulations as compared to the softgel capsule formulation of JNJ-56021927 will be evaluated primarily. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Must agree to use an adequate contraception method as deemed appropriate by the investigator, always use a condom during sexual intercourse, and to not donate sperm during the study and for 3 months after receiving the study drug
* Body mass index between 18 and 30 kilogram (kg) per square meter, and body weight not less than 50 kg
* Blood pressure (supine for 5 minutes) between 90 and 140 millimeter of mercury (mm Hg) systolic, and no higher than 90 mm Hg diastolic
* A 12-lead electrocardiogram (ECG) consistent with normal cardiac conduction and function, including pulse rate between 45 and 99 beats per minute (bpm), QT corrected Fridericia (QTcF) interval less than or equal to 450 milliseconds (msec), QRS interval of less than 120 msec, PR interval less than 220 msec, morphology consistent with healthy cardiac conduction and function
* Nonsmoker within the previous 2 months

Exclusion Criteria:

* History of or current clinically significant medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease, hematologic disease, coagulation disorders (including any abnormal bleeding or blood dyscrasias), lipid abnormalities, significant pulmonary disease, including bronchospastic respiratory disease, diabetes mellitus, hepatic or renal insufficiency, thyroid disease, neurologic or psychiatric disease, infection
* Known hypersensitivity to Vitamin E
* History of stomach or intestinal surgery or resection that would potentially alter absorption or excretion of orally administered drugs
* Known allergy to the study drug or any of the excipients of the formulation
* Unable to swallow solid, oral dosage forms whole with the aid of water

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2014-06; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Maximum Plasma Concentration (Cmax) | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12 , 24, 48, 72, 96, 120, 144, 168, 336, 504, 672, 840, 1008, 1176, 1344 hours post-administration of drug on Day 1
  The Cmax is the maximum observed plasma concentration.
Time to Reach Maximum Concentration (Tmax) | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12 , 24, 48, 72, 96, 120, 144, 168, 336, 504, 672, 840, 1008, 1176, 1344 hours post-administration of drug on Day 1
  The Tmax is time to reach the maximum observed plasma concentration.
Area Under the Plasma Concentration-Time Curve From Time Zero to Time 72 Hours (AUC [0-72]) | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12 , 24, 48, 72 hours post-administration of drug on Day 1
  Area Under the Plasma Concentration-Time Curve From Time Zero to Time 72 Hours (AUC [0-72]) will be evaluated.
Area Under the Plasma Concentration-Time Curve From Time Zero to Time 168 Hours (AUC [0-168]) | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12 , 24, 48, 72, 96, 120, 144, 168 hours post-administration of drug on Day 1
  Area Under the Plasma Concentration-Time Curve From Time Zero to Time 168 Hours (AUC [0-168]) will be evaluated.
Area Under the Plasma Concentration-Time Curve From Time Zero to Last Quantifiable Time (AUC [0-last]) | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12 , 24, 48, 72, 96, 120, 144, 168, 336, 504, 672, 840, 1008, 1176, 1344 hours post-administration of drug on Day 1
  Area under the plasma concentration-time curve from time zero to time of last quantifiable concentration (AUC [0-last]) will be evaluated.
Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0-infinity)] | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12 , 24, 48, 72, 96, 120, 144, 168, 336, 504, 672, 840, 1008, 1176, 1344 hours post-administration of drug on Day 1
  The AUC (0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time, calculated as the sum of AUC (0-last) and Clast/lambda(z), wherein AUC (0-last) is area under the plasma concentration-time curve from time zero to last quantifiable time; Clast is the last observed quantifiable concentration; and lambda(z) is elimination rate constant.
Extrapolated Area Under the Curve (AUC Percent [%] Extrap) | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12 , 24, 48, 72, 96, 120, 144, 168, 336, 504, 672, 840, 1008, 1176, 1344 hours post-administration of drug on Day 1
  The AUC%extrap is the percentage of AUC [0-infinity] obtained by forward extrapolation. It is calculated as (AUC [0-infinity] minus AUC [0-last])*100/ AUC [0-infinity], where AUC [0-infinity] = Area under the plasma concentration versus time curve from time zero (pre-dose) to extrapolated infinite time and AUClast is area under the plasma concentration time-curve from zero (pre-dose) to the last measured concentration.
Elimination Half-Life (t1/2) | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12 , 24, 48, 72, 96, 120, 144, 168, 336, 504, 672, 840, 1008, 1176, 1344 hours post-administration of drug on Day 1
  Elimination half-life (t1/2) is the time measured for the plasma concentration to decrease by one half. Elimination half-life associated with the terminal slope of the semi-logarithmic drug concentration-time curve, calculated as 0.693/elimination rate constant (lambda[z]).
Elimination Rate Constant (lambda[z]) | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12 , 24, 48, 72, 96, 120, 144, 168, 336, 504, 672, 840, 1008, 1176, 1344 hours post-administration of drug on Day 1
  Elimination rate constant is the fraction of a drug that is removed from the body per unit time.
Time to Last Quantifiable Plasma Concentration (Tlast) | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12 , 24, 48, 72, 96, 120, 144, 168, 336, 504, 672, 840, 1008, 1176, 1344 hours post-administration of drug on Day 1
  The Tlast is time to reach the last quantifiable plasma concentration.
Relative Bioavailability | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12 , 24, 48, 72, 96, 120, 144, 168, 336, 504, 672, 840, 1008, 1176, 1344 hours post-administration of drug on Day 1
  Bioavailability means the extent to which the active ingredient of a drug dosage form becomes available at the site of drug action or in a biological medium believed to reflect accessibility to a site of action. Relative bioavailability is the percentage of the administered dose that is systemically available, calculated as: (AUC [0-infinity] of test divided by AUC [0-infinity] of reference) multiplied by 100, where the reference treatment is a non-intravenous administration.
Metabolite to Parent Drug Ratio for Maximum Observed Plasma Concentration (MPR Cmax) | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12 , 24, 48, 72, 96, 120, 144, 168, 336, 504, 672, 840, 1008, 1176, 1344 hours post-administration of drug on Day 1
  The (MPR Cmax) is metabolite to parent drug ratio for maximum observed plasma concentration.
Metabolite to Parent Drug Ratio for Area Under the Plasma Concentration-Time Curve From Time 0 to Last Observed Quantifiable Concentration (MPR AUC[0-last]) | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12 , 24, 48, 72, 96, 120, 144, 168, 336, 504, 672, 840, 1008, 1176, 1344 hours post-administration of drug on Day 1
  The MPR AUClast is metabolite to parent drug ratio for area under the plasma concentration-time curve from time 0 to last quantifiable concentration (AUC [0-last]).
Metabolite to Parent Drug Ratio for Area Under the Plasma Concentration-Time Curve From Time Zero to Extrapolated Infinite Time (MPR AUC [0-infinity]) | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12 , 24, 48, 72, 96, 120, 144, 168, 336, 504, 672, 840, 1008, 1176, 1344 hours post-administration of drug on Day 1
  The MPR AUC [0-infinity] is metabolite to parent drug ratio for area under the plasma concentration-time curve from time zero to extrapolated infinite time (AUC [0-infinity]).

SECONDARY OUTCOMES:
Number of Participants With Treatment-Emergent Adverse Events (AEs) or Serious Adverse Events (SAEs) | Screening up to Day 57 or early withdrawal
  An AE is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to day 57, that are absent before treatment or that worsened relative to pretreatment state.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC